CLINICAL TRIAL: NCT03277937
Title: The Use of Angiography for Determination and Confirmation of the Feeder Vessel as a Modification of the Original EUS-guided Coils and Cyanoacrylate Therapy for Gastric Varices
Brief Title: Angiography for Evaluation of the Feeder Vessel in EUS-guided Coils and Cyanoacrylate Therapy for Gastric Varices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JULY 20-2017
Record Dates: First submitted 2017-07-18; First posted 2017-09-11 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Gastric Varices
Keywords: gastric varices; endoscopic ultrasound; coils; cyanoacrylate
MeSH Terms: conditions — Esophageal and Gastric Varices | interventions — Cyanoacrylates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with gastric varices (Experimental): Patients above 18 years old with gastric varices (GV) on the initial standard diagnostic upper endoscopy will be enrolled and treated using angiography in EUS-injection of coils + CYA. GV will be classified according to Sarin and Kumar classification. Only gastro-esophageal varices type II (GOV II) (fundal varices communicating with esophageal varices) and isolated gastric varices type I (IGV I) (fundal varices within a few centimeters of the gastric cardia) will be included. Gastro-esophageal varices type I (GOV I) will be excluded. Patients with active bleeding and history of previous bleeding due to GV (secondary prophylaxis) will be included as well as patients with high-risk GV suitable for primary prophylaxis according to Baveno VI consensus. T
  Interventions: Procedure: angiography in EUS-injection of coils + CYA

INTERVENTIONS:
Procedure: angiography in EUS-injection of coils + CYA — Doppler imaging will be used to allow direct visualization of the varices flow. The gastric vessels will be followed from the cardia to the proximal part of the esophagus, to detect the feeding vessel (FV). Once the FV has been found, a 19-gauge EUS-FNA will be used to access the vessel. An angiography will be performed using 5-10 ml of water-soluble contrast under fluoroscopy, to ensure intravascular location and study varix flow direction. Finally, patients will be treated by EUS-deployment of coils followed by CYA injection. The coils will be delivered into the vessel through the FNA needle, using the stylet as a pusher. The 2-Octyl-CYA will be used. It will be injected always after the coils deployment and then 1 mL of saline solution will be used to flush the glue completely.
  Other Names: Drug: cyanoacrylate; Device: coils

SUMMARY:
INTRODUCTION: Bleeding from gastric varices (GV) is associated with a high mortality rate. Injection of cyanoacrylate (CYA) using standard gastroscope has demonstrated to achieve higher hemostasis and lower rebleeding rates compared to band ligation or sclerotherapy. Nevertheless CYA treatment is known to be associated with significant adverse events. Pulmonary embolism due to CYA injection is a serious and sometimes fatal complication of this therapy. These patients usually have respiratory symptom, however this complication can be present in asymptomatic patients, being demonstrated only by a pathological CT scan. On the other hand, it has been described that the risk of glue embolism dependent on the volume of CYA injected, being significantly greater with high volumes. Other complications related to CYA injection are hemorrhage from injection site ulcers, fever, peritonitis, needle impaction, and even death. Also the injection material can cause serious damage to the endoscope.

Currently, endoscopic injection of CYA can be performed by direct visualization using a standard gastroscope or guided by Endoscopic Ultrasound (EUS) with injection of CYA alone or in combination with coils. The injection of coils in conjunction with CYA may reduce or eliminate the risk of glue embolization as coils can function as a scaffold to retain CYA within the varix and may decrease the amount of glue injection needed to achieve obliteration. It has been previously demonstrated that treatment under EUS guidance may have some benefits. It allows a precise targeting of the varix lumen or afferent feeding veins, being the vessel obstructed with less amount of CYA than used for the "blind" injection by standard endoscopy, reducing the risk of glue embolism. EUS can confirm varix obliteration by Doppler effect and also the visualization of GV is not impaired by blood or food in the stomach, thus it can be used in the setting of active hemorrhage.

DETAILED DESCRIPTION:
On the other hand, despite the EUS-injection of coils and CYA have shown very promising results, it is extremely important to have experience performing this technique, as the injection in a wrong vessel could be catastrophic. It has been develop in our unit a modification of Binmoeller´s original technique by performing the injection of coils and CYA by EUS and fluoroscopic guidance. The performance of an angiography guided by EUS and under fluoroscopy evaluation, represents a modification to the original technique that add some benefits: 1) The injection of water-soluble contrast allows identifying the variceal flow and the afferent feeding vessel (left gastric vein) and avoiding splenic vessels embolization. 2) Also, if there is a shunt it can be detected and the injection of CYA can be avoided. 3) In case of active bleeding the angiography allows visualizing which varix is bleeding, and target the correct vessel.

The aim of this study is to show the results and potential benefits by adding an angiography to the original EUS-guided injection of coils in combination with CYA technique, to determinate and confirm the feeder vessel in GV treatment.

MATERIALS AND METHODS

Study design: It will be an interventional, descriptive and prospective study, performed in the Ecuadorian Institute of Digestive Disease (IECED), Omni Hospital Academic Tertiary Center Ecuador. Patients have been included from July 2015 and will continue to be included up to October 2017. The study protocol and consent form has been approved by the institutional review board, and will be conducted according to the declaration of Helsinki. Written informed consent will be obtained from all subjects.

Population selection, inclusion and exclusion criteria: Patients above 18 years old with gastric varices (GV) on the initial standard diagnostic upper endoscopy will be enrolled. GV will be classified according to Sarin and Kumar classification. Only gastro-esophageal varices type II (GOV II) (fundal varices communicating with esophageal varices) and isolated gastric varices type I (IGV I) (fundal varices within a few centimeters of the gastric cardia) will be included. Gastro-esophageal varices type I (GOV I) will be excluded as they can be successfully treated by endoscopic band ligation. Patients with active bleeding and history of previous bleeding due to GV (secondary prophylaxis) will be included as well as patients with high-risk GV suitable for primary prophylaxis according to Baveno VI consensus. The exclusion criteria will be pregnancy, concurrent hepatorenal syndrome and/or multi-organ failure, platelet count less than 50,000/ml or International Normalized Rate (INR) >2, esophageal stricture, splenic or portal vein thrombosis and allergy to iodine.

Endoscopic Procedure and Technique: All procedures will be performed in a hospital-based interventional endoscopy setting, where radiology is available and by one endoscopist (C.R.M), under general anesthesia, with tracheal intubation, with the patient in supine position and using antibiotic prophylaxis. EUS examination will be performed using a 3.8 mm working channel linear-array therapeutic echoendoscopes (EG 3870UTK; Pentax, Hamburg, Germany), attached to an ultrasound console (Avius Hitachi, Tokyo, Japan). The echoendoscope will be positioned in the distal esophagus at the level of the cardia (anterograde trans-esophageal, transcrural approach) to visualize the gastric fundus and intramural varices.

Detection of the feeder vessel by EUS: Once positioned, water will be instilled to fill the gastric fundus, in order to improve acoustic coupling and visualization of GV. EUS color Doppler imaging will be used to allow direct visualization of the varices flow. Following the gastric vessel, and by using the fine-flow doppler color of the ultrasound console, the vessel or vessels will be followed from the cardia (distal part of the esophagus) to the proximal part of the esophagus (2 to 3 cm) above the cardia, to detect the feeding vessel. The feeding vessel is characterized by the convergence of all vessels. Once the feeding vessel has been found, a 19 gauge EUS-fine needle aspiration (FNA) (Expect® flexible; Boston Scientific®, Marlborough, USA) will be used to access the vessel, the stylet will be withdrawn and a 20 ml syringe with negative pressure will be used to evaluate blood return, confirming intravascular location. In order to prevent blood clotting of the needle tip, 5 ml of saline solution will be instilled. Moreover, the flush with saline solution allows to confirm the flow of the gastric vessels under B-mode ultrasound visualization.

Using angiography to confirm the target vessel (feeder vessel) and flow traject: In the final diagnostic step, an angiography will be performed using 5 to 10 mL of water-soluble contrast (Ultravist, Bayer, Ecuador) under fluoroscopic evaluation, in order to ensure intravascular location and study varix flow direction (afferent or efferent). Angiography technical success will be measured, determined as the possibility to define the flow trajectory vessel under fluoroscopy.

EUS-guided deployment of Coils and Cyanoacrylate injection: Finally, patients will be treated by EUS-deployment of coils followed by CYA injection. The intravascular embolization coils that will be used (10-16 mm coiled diameter, 12-20 cm straight lengths, 0.035 inches diameter, Nester Embolization Coil; Cook Medical) will be delivered into the vessel through the FNA needle, using the stylet as a pusher. Special attention will be paid not place the needle tip on the counter wall due to the risk of perforation, bleed, coil extrusion and to allow enough space for the coil to curl.

The CYA that will be used is the 2-Octyl-CYA (Dermabond; Ethicon, Piscataway, NJ). It will be injected always after the coils are deployed and then 1 mL of saline solution will be used to flush the glue completely through the needle. The diameter (10-16 mm), number of coils and the volume of the 2-Octyl-CYA injected will be calculated according to the diameter of the vessel measured on EUS and by the angiography of the vessel. After 30 seconds, once CYA has been solidified and the risk of bleeding on the puncturing site decrease, the needle will be withdrawn. Obliteration of the vessel will be confirmed 3 minutes later using Doppler imaging. Complete obliteration of the treated varix will be defined as absence of Doppler flow on EUS.

A direct visualization of the gastric varices will be performed after the EUS procedure to determine the effect of the obliteration of the feeder vessel by using a standard videoendoscope. After the procedure, patients will be observed for 2 hours in the recovery room before being discharged of the unit. In cases of primary prophylaxis the treatment will be ambulatory.

Finally, a 1, 3, 9 and 12 months follow-up will be performed in order to confirm the results of the EUS-therapeutic by EUS and by upper endoscopy.

Technical success will be considered as target of the vessels and deployment of the proposed EUS-therapeutic. Treatment failure and early rebleeding will be considered when bleeding occurred the first five days and between 5 and 90 days respectively.

Statistical analysis: Demographic characteristics, previous medication and radiological images will be described. Quantitative variables will be described in mean or median, and standard deviation or range, as corresponding. Qualitative variables will be described in percentages. A Kolmogorov-Smirnov test with a p value <0.05 will be considered to be statistically significant. The IECED institutional biostatistician will review statistical methodology of the study. Statistical calculations will be performed in SPSS software suite v.22.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years old with gastric varices (GV) on the initial standard diagnostic upper endoscopy will be enrolled. GV will be classified
* Only gastro-esophageal varices type II (GOV II) (fundal varices communicating with esophageal varices) and isolated gastric varices type I (IGV I) (fundal varices within a few centimeters of the gastric cardia) will be included (according to Sarin and Kumar classification).
* Patients with active bleeding and history of previous bleeding due to GV (secondary prophylaxis)
* Patients with high-risk GV suitable for primary prophylaxis according to Baveno VI consensus.

Exclusion Criteria:

* Gastro-esophageal varices type I (GOV I) will be excluded as they can be successfully treated by endoscopic band ligation.
* Pregnancy,
* Hepatorenal syndrome
* Multi-organ failure,
* platelet count less than 50,000/ml
* International Normalized Rate (INR) >2,
* esophageal stricture,
* Splenic vein thrombosis
* Portal vein thrombosis
* Allergy to iodine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
efficacy of adding angiography to the EUS-guided injection of coils + CYA technique, to determinate, confirm and target the feeder vessel in GV treatment. | 12 months
  efficacy will be considered be the complete occlusion and/or disappearance of the GV and will be determinate by follow-up controls using EUS and upper endoscopy. Treatment failure and early rebleeding will be considered when bleeding occurred the first five days.

SECONDARY OUTCOMES:
safety of adding angiography to the EUS-guided injection of coils + CYA technique, to determinate and confirm the feeder vessel in GV treatment | 12 months
  all adverse events related to the technique during the procedure or the follow-up will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Robles-Medranda, MD, Principal Investigator — Ecuadorian Institute of Digestive Diseases
Locations (1):
- Ecuadorian Institute of Digestive Diseases, Omnihospital, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hashizume M, Akahoshi T, Tomikawa M. Management of gastric varices. J Gastroenterol Hepatol. 2011 Jan;26 Suppl 1:102-8. doi: 10.1111/j.1440-1746.2010.06572.x. PMID 21199520
- [Result] Sarin SK, Sachdev G, Nanda R, Misra SP, Broor SL. Endoscopic sclerotherapy in the treatment of gastric varices. Br J Surg. 1988 Aug;75(8):747-50. doi: 10.1002/bjs.1800750809. PMID 3262398
- [Result] Irani S, Kowdley K, Kozarek R. Gastric varices: an updated review of management. J Clin Gastroenterol. 2011 Feb;45(2):133-48. doi: 10.1097/MCG.0b013e3181fbe249. PMID 21135706
- [Result] Mahadeva S, Bellamy MC, Kessel D, Davies MH, Millson CE. Cost-effectiveness of N-butyl-2-cyanoacrylate (histoacryl) glue injections versus transjugular intrahepatic portosystemic shunt in the management of acute gastric variceal bleeding. Am J Gastroenterol. 2003 Dec;98(12):2688-93. doi: 10.1111/j.1572-0241.2003.08769.x. PMID 14687818
- [Result] Cheng LF, Wang ZQ, Li CZ, Cai FC, Huang QY, Linghu EQ, Li W, Chai GJ, Sun GH, Mao YP, Wang YM, Li J, Gao P, Fan TY. Treatment of gastric varices by endoscopic sclerotherapy using butyl cyanoacrylate: 10 years' experience of 635 cases. Chin Med J (Engl). 2007 Dec 5;120(23):2081-5. PMID 18167180
- [Result] Seewald S, Ang TL, Imazu H, Naga M, Omar S, Groth S, Seitz U, Zhong Y, Thonke F, Soehendra N. A standardized injection technique and regimen ensures success and safety of N-butyl-2-cyanoacrylate injection for the treatment of gastric fundal varices (with videos). Gastrointest Endosc. 2008 Sep;68(3):447-54. doi: 10.1016/j.gie.2008.02.050. PMID 18760173
- [Result] Romero-Castro R, Ellrichmann M, Ortiz-Moyano C, Subtil-Inigo JC, Junquera-Florez F, Gornals JB, Repiso-Ortega A, Vila-Costas J, Marcos-Sanchez F, Munoz-Navas M, Romero-Gomez M, Brullet-Benedi E, Romero-Vazquez J, Caunedo-Alvarez A, Pellicer-Bautista F, Herrerias-Gutierrez JM, Fritscher-Ravens A. EUS-guided coil versus cyanoacrylate therapy for the treatment of gastric varices: a multicenter study (with videos). Gastrointest Endosc. 2013 Nov;78(5):711-21. doi: 10.1016/j.gie.2013.05.009. Epub 2013 Jul 25. PMID 23891417
- [Result] Hwang SS, Kim HH, Park SH, Kim SE, Jung JI, Ahn BY, Kim SH, Chung SK, Park YH, Choi KH. N-butyl-2-cyanoacrylate pulmonary embolism after endoscopic injection sclerotherapy for gastric variceal bleeding. J Comput Assist Tomogr. 2001 Jan-Feb;25(1):16-22. doi: 10.1097/00004728-200101000-00003. PMID 11176287
- [Result] Kok K, Bond RP, Duncan IC, Fourie PA, Ziady C, van den Bogaerde JB, van der Merwe SW. Distal embolization and local vessel wall ulceration after gastric variceal obliteration with N-butyl-2-cyanoacrylate: a case report and review of the literature. Endoscopy. 2004 May;36(5):442-6. doi: 10.1055/s-2004-814323. PMID 15100955
- [Result] Sarin SK, Jain AK, Jain M, Gupta R. A randomized controlled trial of cyanoacrylate versus alcohol injection in patients with isolated fundic varices. Am J Gastroenterol. 2002 Apr;97(4):1010-5. doi: 10.1111/j.1572-0241.2002.05622.x. PMID 12003381
- [Result] Noophun P, Kongkam P, Gonlachanvit S, Rerknimitr R. Bleeding gastric varices: results of endoscopic injection with cyanoacrylate at King Chulalongkorn Memorial Hospital. World J Gastroenterol. 2005 Dec 21;11(47):7531-5. doi: 10.3748/wjg.v11.i47.7531. PMID 16437729
- [Result] Bhasin DK, Sharma BC, Prasad H, Singh K. Endoscopic removal of sclerotherapy needle from gastric varix after N-butyl-2-cyanoacrylate injection. Gastrointest Endosc. 2000 Apr;51(4 Pt 1):497-8. doi: 10.1016/s0016-5107(00)70459-7. No abstract available. PMID 10744834
- [Result] Saracco G, Giordanino C, Roberto N, Ezio D, Luca T, Caronna S, Carucci P, De Bernardi Venon W, Barletti C, Bruno M, De Angelis C, Musso A, Repici A, Suriani R, Rizzetto M. Fatal multiple systemic embolisms after injection of cyanoacrylate in bleeding gastric varices of a patient who was noncirrhotic but with idiopathic portal hypertension. Gastrointest Endosc. 2007 Feb;65(2):345-7. doi: 10.1016/j.gie.2006.07.009. Epub 2006 Dec 1. No abstract available. PMID 17141231
- [Result] Rickman OB, Utz JP, Aughenbaugh GL, Gostout CJ. Pulmonary embolization of 2-octyl cyanoacrylate after endoscopic injection therapy for gastric variceal bleeding. Mayo Clin Proc. 2004 Nov;79(11):1455-8. doi: 10.4065/79.11.1455. PMID 15544027
- [Result] Bhat YM, Weilert F, Fredrick RT, Kane SD, Shah JN, Hamerski CM, Binmoeller KF. EUS-guided treatment of gastric fundal varices with combined injection of coils and cyanoacrylate glue: a large U.S. experience over 6 years (with video). Gastrointest Endosc. 2016 Jun;83(6):1164-72. doi: 10.1016/j.gie.2015.09.040. Epub 2015 Oct 9. PMID 26452992
- [Result] Romero-Castro R, Pellicer-Bautista F, Giovannini M, Marcos-Sanchez F, Caparros-Escudero C, Jimenez-Saenz M, Gomez-Parra M, Arenzana-Seisdedos A, Leria-Yebenes V, Herrerias-Gutierrez JM. Endoscopic ultrasound (EUS)-guided coil embolization therapy in gastric varices. Endoscopy. 2010;42 Suppl 2:E35-6. doi: 10.1055/s-0029-1215261. Epub 2010 Jan 13. No abstract available. PMID 20073010
- [Result] Iwase H, Suga S, Morise K, Kuroiwa A, Yamaguchi T, Horiuchi Y. Color Doppler endoscopic ultrasonography for the evaluation of gastric varices and endoscopic obliteration with cyanoacrylate glue. Gastrointest Endosc. 1995 Feb;41(2):150-4. doi: 10.1016/s0016-5107(05)80599-1. No abstract available. PMID 7721004
- [Result] Levy MJ, Wong Kee Song LM, Kendrick ML, Misra S, Gostout CJ. EUS-guided coil embolization for refractory ectopic variceal bleeding (with videos). Gastrointest Endosc. 2008 Mar;67(3):572-4. doi: 10.1016/j.gie.2007.06.063. Epub 2007 Nov 12. No abstract available. PMID 17997404
- [Result] Lee YT, Chan FK, Ng EK, Leung VK, Law KB, Yung MY, Chung SC, Sung JJ. EUS-guided injection of cyanoacrylate for bleeding gastric varices. Gastrointest Endosc. 2000 Aug;52(2):168-74. doi: 10.1067/mge.2000.107911. PMID 10922086
- [Result] Romero-Castro R, Pellicer-Bautista FJ, Jimenez-Saenz M, Marcos-Sanchez F, Caunedo-Alvarez A, Ortiz-Moyano C, Gomez-Parra M, Herrerias-Gutierrez JM. EUS-guided injection of cyanoacrylate in perforating feeding veins in gastric varices: results in 5 cases. Gastrointest Endosc. 2007 Aug;66(2):402-7. doi: 10.1016/j.gie.2007.03.008. PMID 17643723
- [Result] Gubler C, Bauerfeind P. Safe and successful endoscopic initial treatment and long-term eradication of gastric varices by endoscopic ultrasound-guided Histoacryl (N-butyl-2-cyanoacrylate) injection. Scand J Gastroenterol. 2014 Sep;49(9):1136-42. doi: 10.3109/00365521.2014.929171. Epub 2014 Jun 20. PMID 24947448
- [Result] Fujii-Lau LL, Law R, Wong Kee Song LM, Gostout CJ, Kamath PS, Levy MJ. Endoscopic ultrasound (EUS)-guided coil injection therapy of esophagogastric and ectopic varices. Surg Endosc. 2016 Apr;30(4):1396-404. doi: 10.1007/s00464-015-4342-3. Epub 2015 Jul 3. PMID 26139494
- [Result] Binmoeller KF, Weilert F, Shah JN, Kim J. EUS-guided transesophageal treatment of gastric fundal varices with combined coiling and cyanoacrylate glue injection (with videos). Gastrointest Endosc. 2011 Nov;74(5):1019-25. doi: 10.1016/j.gie.2011.06.030. Epub 2011 Sep 1. PMID 21889139
- [Result] Sarin SK, Kumar A. Gastric varices: profile, classification, and management. Am J Gastroenterol. 1989 Oct;84(10):1244-9. PMID 2679046
- [Result] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Result] Gianotti R, Charles H, Hymes K, Chandarana H, Sigal S. Treatment of gastric varices with partial splenic embolization in a patient with portal vein thrombosis and a myeloproliferative disorder. World J Gastroenterol. 2014 Oct 21;20(39):14495-9. doi: 10.3748/wjg.v20.i39.14495. PMID 25339837
- [Result] Rengstorff DS, Binmoeller KF. A pilot study of 2-octyl cyanoacrylate injection for treatment of gastric fundal varices in humans. Gastrointest Endosc. 2004 Apr;59(4):553-8. doi: 10.1016/s0016-5107(03)02865-7. PMID 15044898